CLINICAL TRIAL: NCT04111094
Title: Urinary Dickkopf-3 for Prognosis and Monitoring of Glomerular Filtration Rate Decline in Patients With Heart Failure
Brief Title: DKK3 for Prognosis and Monitoring of GFR Decline in Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 122/19
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HF: Diagnosed heart failure as described by recent guidelines. Inclusion criteria will be applied: i) minimum one symptom typical of HF: positive physical examination (e.g., bilateral oedema, increased jugular pressure) or positive clinical history (e.g., orthopnoea, history of coronary vascular disease, history of arterial hypertension, exposition to cardiotoxic drug/radiation, diuretic use); b-type natriuretic peptide (BNP) or N-terminal pro-BNP levels ≥35 or ≥125 pg/ml, respectively; and iii) classification as New York Heart Association (NYHA) functional class 2 or 3. There is no prespecified inclusion criterion with respect to left ventricular ejection fraction as congestive symptoms and prevalence of kidney dysfunction are comparable in patients with HF across the left ventricular ejection fraction spectrum.
  Interventions: Diagnostic Test: No intervention
- Diabetes mellitus/hypertension: Diagnosed diabetes mellitus, with/without treatment
  Interventions: Diagnostic Test: No intervention
- Hypertension: Diagnosed hypertension, with/without treatment
  Interventions: Diagnostic Test: No intervention
- Cystic kidney diseases: Diagnosed cystic kidney diseases, with/without treatment
  Interventions: Diagnostic Test: No intervention
- Tubulointerstitial diseases: Diagnosed tubulointerstitial diseases, with/without treatment
  Interventions: Diagnostic Test: No intervention
- Glomerular diseases: Diagnosed glomerular diseases, with/without treatment
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
The individual course of chronic kidney disease (CKD) may vary, and improved methods for identifying which patients will experience estimated glomerular filtration rate (eGFR) decline are needed. Recently, urinary dickkopf-3 (DKK3) has been proposed to predict eGFR decline in patients with CKD, independent of presence of albuminuria. The investigators sought to examine the association between changes in DKK3 levels and eGFR decline in patients with heart failure (HF).

DETAILED DESCRIPTION:
The individual course of chronic kidney disease (CKD) may vary, and improved methods for identifying which patients will experience estimated glomerular filtration rate (eGFR) decline are needed. Recently, urinary dickkopf-3 (DKK3) has been identified as an stress-induced, renal tubular epithelia-derived, secreted glycoprotein that induces tubulointerstitial fibrosis. Urinary DKK3 has been found to predict eGFR decline in patients with CKD, independent of presence of albuminuria, but its association with eGFR decline in patients with heart failure (HF) is unknown. The investigators sought to examine the association between changes in DKK3 and eGFR decline in patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥18 years of age with diagnosed HF or diabetes or hypertension

Exclusion Criteria:

* CKD with estimated GFR <20 ml/min/1.73 m2 (2012 CKD-EPI equation)
* CKD with extracorporeal or peritoneal ultrafiltration due to diuretic-resistant fluid overload
* active tumor disease
* inflammatory or autoimmune disease requiring systemic immunosuppressive treatment
* clinically apparent infections
* recipients of solid-organ transplants
* anticipated life expectancy of <12 months
* likelihood of receiving advanced therapy (mechanical circulatory assist device/cardiac transplant)
* pregnancy or possibility of pregnancy in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients ≥18 years of age with diagnosed HF or diabetes or hypertension or other etiologies of CKD
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Association between DKK3 and eGFR decline | 24 months
  DKK3 and eGFR (CKD-Epidemiology Collaboration equation)

SECONDARY OUTCOMES:
Association between proteinuria and DKK3 | 24 months
  DKK3 and proteinuria, albuminuria, and alpha 1 microglobulin excretion
Persistent or worsening of HF | 24 months
  Cardiovascular death, hospital admission for decompensated HF, or clinical HF decompensation without hospital admission (but requiring parenteral HF therapy or changes in oral HF medications including diuretics)
Need for renal replacement therapy | 24 months
  Requirement of incident renal replacement therapy
Association of venous congestion/volume overload with DKK3 | 24 months
  B-type natriuretic peptide, clinical examination, bioimpedance analysis, echocardiography
Association of right and left ventricular function with DKK3 | 24 months
  Echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Chair — University Hospital Giessen
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zewinger S, Rauen T, Rudnicki M, Federico G, Wagner M, Triem S, Schunk SJ, Petrakis I, Schmit D, Wagenpfeil S, Heine GH, Mayer G, Floege J, Fliser D, Grone HJ, Speer T. Dickkopf-3 (DKK3) in Urine Identifies Patients with Short-Term Risk of eGFR Loss. J Am Soc Nephrol. 2018 Nov;29(11):2722-2733. doi: 10.1681/ASN.2018040405. Epub 2018 Oct 2. PMID 30279273
- [Background] Federico G, Meister M, Mathow D, Heine GH, Moldenhauer G, Popovic ZV, Nordstrom V, Kopp-Schneider A, Hielscher T, Nelson PJ, Schaefer F, Porubsky S, Fliser D, Arnold B, Grone HJ. Tubular Dickkopf-3 promotes the development of renal atrophy and fibrosis. JCI Insight. 2016 Jan 21;1(1):e84916. doi: 10.1172/jci.insight.84916. PMID 27699213